CLINICAL TRIAL: NCT01013467
Title: Does a Colour-coded Blood Pressure Diary Improve Blood Pressure Control for Patients in General Practice? A Randomised Controlled Study
Brief Title: CoCo: Colour Coded Blood Pressure Control
Acronym: CoCo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1738
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Hypertension
Keywords: blood pressure; control; adherence; behaviour
MeSH Terms: conditions — Hypertension; Behavior

ARMS (1):
- color coded bloodpressure booklet (Active Comparator)
  Interventions: Behavioral: "CoCo" colour coded blood pressure control

INTERVENTIONS:
Behavioral: "CoCo" colour coded blood pressure control — The patients in the intervention group will receive a colour-coded blood pressure record booklet. The corresponding colour coded areas are divided into three areas of green, yellow and red following a traffic light system. The green area covers blood pressure readings up to a maximum of 140/90 mmHg, the yellow area includes systolic readings over 140 to 180 mm Hg and diastolic readings over 90 to 110 mmHg. The red area covers systolic readings over 180 mmHg and diastolic readings over 110 mmHg.

SUMMARY:
Insufficient blood pressure control is a frequent problem despite the existence of effective treatment. One of the causes is insufficient self-monitoring and a lack of adherence to therapy. Blood pressure self-measurement at home (Home Blood Pressure Measurement, HBPM) has positive effects on treatment adherence and is helpful in achieving the target blood pressure.

Only a few studies have investigated whether the adherence for HBPM can be improved through simple measures and better blood pressure monitoring can be achieved.

Objective Improvement of self-monitoring by means of blood pressure self-measurement and improved blood pressure control by using a new colour-coded blood pressure diary

ELIGIBILITY:
Inclusion criteria:

* Age >18 years
* BP > 140/90 mmHg Two consecutive measurements carried out in the practice (measured by the general practitioner at the start of the study).
* Unchanged anti-hypertension treatment for one month before inclusion
* Patient able to measure blood pressure at home
* Written informed consent

Exclusion criteria: • Blood pressure reading over 180 mmHg systolic and/or 110 mmHg diastolic.

* Serious general or psychological illness (malignant tumor, serious depressive episodes or evidence of dementia).
* Insufficient knowledge of the German language for instruction and blood pressure recording with a booklet.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2009-10; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Primary outcome: change in systolic and/or diastolic blood pressure 6 months after using the new colour-coded blood pressure diary. | 6months

SECONDARY OUTCOMES:
adherence with home blood pressure measurements | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Rosemann, Prof MD, Principal Investigator — University Hospital Zurich, Institute of General Practice
Locations (1):
- University Hospital Zurich, Institute of General Practice, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Steurer-Stey C, Zoller M, Chmiel Moshinsky C, Senn O, Rosemann T. Does a colour-coded blood pressure diary improve blood pressure control for patients in general practice: the CoCo trial. Trials. 2010 Apr 14;11:38. doi: 10.1186/1745-6215-11-38. PMID 20398258